CLINICAL TRIAL: NCT01561482
Title: Open-Label Study Of Metformin In Combination With Simvastatin For Men With Prostate Carcinoma And A Rising Serum Prostate-Specific Antigen Level After Radical Prostatectomy And/Or Radiation Therapy
Brief Title: Study of Metformin With Simvastatin for Men With Prostate Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed due to slow/low enrollment; no subjects were enrolled.
Sponsor: Nicholas Mitsiades (Other)
Responsible Party: Sponsor-Investigator, Nicholas Mitsiades, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28936
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Prostate Carcinoma
Keywords: Prostate carcinoma; Prostate cancer; Prostate Specific Antigen; PSA; Metformin; Simvastatin; Radiation therapy; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin, Simvastatin (Experimental): Both metformin and simvastatin will be taken every day. Metformin will be taken as 1 pill in the morning and 1 pill before going to bed. Simvastatin will be taken as 1 pill before going to bed.
  They will be taken until metastasis from the prostate cancer appears or until the subjects PSA has doubled from what it was before they started the study.
  Interventions: Drug: Metformin; Drug: Simvastatin

INTERVENTIONS:
Drug: Metformin — Metformin treatment will be started at 500 mg twice daily (dose level -2), in order to minimize gastrointestinal discomfort and, if no gastrointestinal toxicity grade greater than 1, will be increased to 500 mg with breakfast/1000 mg at bedtime (dose level -1) 4 days later (+/- 1 day allowed). If no gastrointestinal toxicity grade greater than 1, it will be increased to 1000 mg twice daily (dose level 0) 10 days later (+/- 2 days allowed), which is the target dose for the remainder of the study. If gastrointestinal toxicity grade greater than 1 occurs during these first 4 weeks, the subject will be evaluated every 2 weeks until resolution of toxicity to grade less than or equal to 1 and, then, the metformin dose will be increased to the next dose level.
  Other Names: Glucophage
Drug: Simvastatin — The simvastatin dose at treatment initiation will be 20 mg once daily (dose level -1), taken at bedtime for 2 weeks. After these 2 weeks, the subject will have blood work and, if no AST/ALT/CPK elevation grade greater than 1, will be escalated to 40 mg once daily (dose level 0), taken at bedtime. If AST or ALT or CPK elevation grade greater than 1 during the first 2 weeks, the subject will be evaluated every 2 weeks until resolution of toxicity to grade less than or equal to 1, and then the simvastatin dose will be increased to dose level 0.
  Other Names: Zocor

SUMMARY:
The purpose of this study is to find out whether the two drugs used in the study, metformin and simvastatin, can slow down the speed of rise of prostate specific antigen (PSA) or stop its rise or even bring the level down.

Recently, scientists noticed that men who take metformin to treat their high blood sugar or simvastatin to treat their high cholesterol are less likely to develop prostate cancer. Also, scientists found that, when these drugs are used in preclinical studies, they can slow down the growth of the prostate cancer cells. This study will try to find out whether these drugs can actually slow down the growth of prostate cancer in men.

DETAILED DESCRIPTION:
Men who participate in this study will take both metformin and simvastatin every day. Both drugs are pills and can be taken at home.

Subjects will be asked to take metformin and simvastatin until metastasis from their prostate cancer appears or until their PSA has doubled from what it was before they started the study.

Primary Objective:

To define the efficacy, as measured by an improvement in PSA doubling time (PSADT) at 6 months, of the combination of metformin plus simvastatin in patients with recurrent prostate cancer following definitive treatment.

Secondary Objectives:

1. To define the time to protocol-specified event for men treated with the combination of metformin plus simvastatin.
2. To describe the pattern of change in log PSA levels and PSA velocity over time during treatment with metformin plus simvastatin.
3. To describe the associations between changes in metabolic parameters (fasting glucose/insulin/lipid panel/leptin/adiponectin and others) with the pattern of change in log PSA levels.

ELIGIBILITY:
Inclusion Criteria:

The study population will consist of subjects who have undergone primary therapy (prostatectomy or primary radiation) for biopsy-proven adenocarcinoma of the prostate and now have biochemical-only recurrence.

1. Ability to understand and the willingness to sign a written informed consent document.
2. Male 18 years or older.
3. Histologically or cytologically confirmed diagnosis of prostate cancer.
4. Biochemical recurrence following prostatectomy or radiation to the prostate, defined as at least 3 PSA rises, with each PSA determination at least 4 weeks apart, and each PSA value greater than or equal to 0.2 ng/mL.
5. PSA must be less than 50 ng/mL at study entry.
6. Screening PSA greater than or equal to 0.5 ng/mL for men who had a prostatectomy. Prior treatment with neoadjuvant, adjuvant, or salvage radiation therapy is allowed, again, with screening PSA greater than or equal to 0.5 ng/mL required for eligibility.
7. Screening PSA greater than or equal to 1.0 ng/mL above their postradiation nadir for men who were treated with primary radiation therapy (external beam and/or brachytherapy). Men who had primary radiation therapy followed by salvage prostatectomy are eligible if screening PSA is greater than or equal to 0.5 ng/mL.
8. PSA doubling time between 3 and 36 months.
9. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
10. Subjects must have normal organ and marrow function as defined below:

    * Leukocytes greater than or equal to 3,000/mcL * Absolute neutrophil count greater than or equal to 1,500/mcL * Hemoglobin greater than or equal to 10 g/dL * Platelets greater than or equal to 100,000/mcL * Total bilirubin within normal institutional limits * AST(SGOT)/ALT(SGPT) less than or equal to 1.5 X institutional upper limit of normal * Creatinine within normal institutional limits OR creatinine clearance or calculated greater than or equal to 60 mL/min/1.73 m2 for subjects with creatinine clearance or estimated creatinine levels above institutional glomerular filtration rate (eGFR) normal * Creatine phosphokinase (CPK) less than or equal to the institutional upper limit of normal
11. Ability to swallow the study drugs.
12. Life expectancy of at least 12 months.
13. Subjects should agree to avoid grapefruit juice which is a major inhibitor of CYP3A4.

Exclusion Criteria:

1. Evidence of metastatic disease on imaging studies.
2. Need for treatment with any conventional modality for prostate cancer (surgery, radiation therapy, and hormonal therapy).
3. Prior hormonal therapy for recurrent prostate cancer (hormonal therapy given in a neoadjuvant or adjuvant setting and greater than 6 months before entry is acceptable).
4. Prior chemotherapy for prostate cancer.
5. Treatment within the last 30 days with any investigational drug.
6. Radiation therapy within prior 6 months.
7. Known hypersensitivity to metformin or statins.
8. Subjects who need to take CYP3A4 inhibitors, such as cyclosporin, sirolimus, tacrolimus, verapamil,danazol, gemfibrozil, ketoconazole, or macrolide antibiotics (e.g., azithromycin, clarithromycin, erythromycin)will be excluded. Prior use of these agents is acceptable, as long as they are stopped at least a week prior to study entry.
9. Subjects who need to take CYP3A4 inducers, such as phenobarbital, dexamethasone, carbamazepine,phenytoin, rifampicin, or non-nucleoside reverse transcriptase inhibitors (e.g., efavirenz, nevirapine,etravirine) will be excluded. Prior use of these agents is acceptable, as long as they are stopped at least a week prior to study entry.
10. Prior history of rhabdomyolysis.
11. Prior history of lactic acidosis.
12. Any history of myocardial infarction in the past 12 months.
13. HIV-positive status.
14. Subjects who consume more than 3 alcoholic beverages per day.
15. Subjects with serious intercurrent illness, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or other nonmalignant medical or psychiatric illness that is uncontrolled or whose control may be jeopardized by the complications of this therapy or may limit compliance with the study requirements (at the discretion of the investigator).
16. Subjects diagnosed with or treated for another malignancy within 2 years prior to study enrollment or previously diagnosed with another malignancy and still having any evidence of residual disease. Subjects with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
17. Subjects currently treated with metformin or a statin or who have been treated with metformin or a statin in the past 6 months are ineligible for this study.
18. Subjects who have taken 5a-reductase inhibitors (finasteride or dutasteride), saw palmetto, or PC-SPES within the last 6 weeks are ineligible for this study. Subjects taking other herbal supplements, vitamins, or other alternative medications are eligible for this study as long as they were started more than 2 months prior to study entry, have remained on a stable regimen, and will remain on a stable regimen for the duration of participation on this study.

Men of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Efficacy, as measured by an improvement in PSA doubling time (PSADT) between baseline and 6 months, of the combination of metformin plus simvastatin in patients with recurrent prostate cancer following definitive treatment. | 6 months after subject start of study

SECONDARY OUTCOMES:
Time to protocol-specified event for men treated with the combination of metformin plus simvastatin. | From treatment initiation till disease progression (assessed up to 5 years)
Pattern of change in log PSA levels and PSA velocity over time during treatment with metformin plus simvastatin. | From treatment initiation till disease progression (assessed up to 5 years)
Associations between changes in metabolic parameters (fasting glucose/insulin/lipid panel/leptin/adiponectin and others) with the pattern of change in log PSA levels. | From treatment initiation till disease progression (assessed up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Mitsiades, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E. Debakey Veterans Affairs Medical Center, Houston, Texas

REFERENCES:
- [Background] Bonorden MJ, Rogozina OP, Kluczny CM, Grossmann ME, Grambsch PL, Grande JP, Perkins S, Lokshin A, Cleary MP. Intermittent calorie restriction delays prostate tumor detection and increases survival time in TRAMP mice. Nutr Cancer. 2009;61(2):265-75. doi: 10.1080/01635580802419798. PMID 19235043
- [Background] Giovanella BC, Shepard RC, Stehlin JS, Venditti JM, Abbott BJ. Calorie restriction: effect on growth of human tumors heterotransplanted in nude mice. J Natl Cancer Inst. 1982 Feb;68(2):249-57. PMID 6278189
- [Background] Hermann LS. Metformin: a review of its pharmacological properties and therapeutic use. Diabete Metab. 1979 Sep;5(3):233-45. PMID 387488
- [Background] Sarkar NH, Fernandes G, Telang NT, Kourides IA, Good RA. Low-calorie diet prevents the development of mammary tumors in C3H mice and reduces circulating prolactin level, murine mammary tumor virus expression, and proliferation of mammary alveolar cells. Proc Natl Acad Sci U S A. 1982 Dec;79(24):7758-62. doi: 10.1073/pnas.79.24.7758. PMID 6296850
- [Background] Albanes D. Caloric intake, body weight, and cancer: a review. Nutr Cancer. 1987;9(4):199-217. doi: 10.1080/01635588709513929. PMID 3299283
- [Background] Bailey CJ. Biguanides and NIDDM. Diabetes Care. 1992 Jun;15(6):755-72. doi: 10.2337/diacare.15.6.755. PMID 1600835
- [Background] Hursting SD, Switzer BR, French JE, Kari FW. The growth hormone: insulin-like growth factor 1 axis is a mediator of diet restriction-induced inhibition of mononuclear cell leukemia in Fischer rats. Cancer Res. 1993 Jun 15;53(12):2750-7. PMID 8389243
- [Background] Frederich RC, Hamann A, Anderson S, Lollmann B, Lowell BB, Flier JS. Leptin levels reflect body lipid content in mice: evidence for diet-induced resistance to leptin action. Nat Med. 1995 Dec;1(12):1311-4. doi: 10.1038/nm1295-1311. PMID 7489415
- [Background] Frederich RC, Lollmann B, Hamann A, Napolitano-Rosen A, Kahn BB, Lowell BB, Flier JS. Expression of ob mRNA and its encoded protein in rodents. Impact of nutrition and obesity. J Clin Invest. 1995 Sep;96(3):1658-63. doi: 10.1172/JCI118206. PMID 7657836
- [Background] Frystyk J, Vestbo E, Skjaerbaek C, Mogensen CE, Orskov H. Free insulin-like growth factors in human obesity. Metabolism. 1995 Oct;44(10 Suppl 4):37-44. doi: 10.1016/0026-0495(95)90219-8. PMID 7476310
- [Background] Halaas JL, Gajiwala KS, Maffei M, Cohen SL, Chait BT, Rabinowitz D, Lallone RL, Burley SK, Friedman JM. Weight-reducing effects of the plasma protein encoded by the obese gene. Science. 1995 Jul 28;269(5223):543-6. doi: 10.1126/science.7624777.
- [Background] Scherer PE, Williams S, Fogliano M, Baldini G, Lodish HF. A novel serum protein similar to C1q, produced exclusively in adipocytes. J Biol Chem. 1995 Nov 10;270(45):26746-9. doi: 10.1074/jbc.270.45.26746. PMID 7592907
- [Background] Burfeind P, Chernicky CL, Rininsland F, Ilan J, Ilan J. Antisense RNA to the type I insulin-like growth factor receptor suppresses tumor growth and prevents invasion by rat prostate cancer cells in vivo. Proc Natl Acad Sci U S A. 1996 Jul 9;93(14):7263-8. doi: 10.1073/pnas.93.14.7263. PMID 8692980
- [Background] Cioffi JA, Shafer AW, Zupancic TJ, Smith-Gbur J, Mikhail A, Platika D, Snodgrass HR. Novel B219/OB receptor isoforms: possible role of leptin in hematopoiesis and reproduction. Nat Med. 1996 May;2(5):585-9. doi: 10.1038/nm0596-585. PMID 8616721
- [Background] Considine RV, Sinha MK, Heiman ML, Kriauciunas A, Stephens TW, Nyce MR, Ohannesian JP, Marco CC, McKee LJ, Bauer TL, et al. Serum immunoreactive-leptin concentrations in normal-weight and obese humans. N Engl J Med. 1996 Feb 1;334(5):292-5. doi: 10.1056/NEJM199602013340503. PMID 8532024
- [Background] Hu E, Liang P, Spiegelman BM. AdipoQ is a novel adipose-specific gene dysregulated in obesity. J Biol Chem. 1996 May 3;271(18):10697-703. doi: 10.1074/jbc.271.18.10697. PMID 8631877
- [Background] Spiegelman BM, Flier JS. Adipogenesis and obesity: rounding out the big picture. Cell. 1996 Nov 1;87(3):377-89. doi: 10.1016/s0092-8674(00)81359-8. No abstract available. PMID 8898192
- [Background] Andersson SO, Wolk A, Bergstrom R, Adami HO, Engholm G, Englund A, Nyren O. Body size and prostate cancer: a 20-year follow-up study among 135006 Swedish construction workers. J Natl Cancer Inst. 1997 Mar 5;89(5):385-9. doi: 10.1093/jnci/89.5.385. PMID 9060961
- [Background] Dunn SE, Kari FW, French J, Leininger JR, Travlos G, Wilson R, Barrett JC. Dietary restriction reduces insulin-like growth factor I levels, which modulates apoptosis, cell proliferation, and tumor progression in p53-deficient mice. Cancer Res. 1997 Nov 1;57(21):4667-72. PMID 9354418
- [Background] Blum WF, Englaro P, Attanasio AM, Kiess W, Rascher W. Human and clinical perspectives on leptin. Proc Nutr Soc. 1998 Aug;57(3):477-85. doi: 10.1079/pns19980068. No abstract available. PMID 9794007
- [Background] Hankinson SE, Willett WC, Colditz GA, Hunter DJ, Michaud DS, Deroo B, Rosner B, Speizer FE, Pollak M. Circulating concentrations of insulin-like growth factor-I and risk of breast cancer. Lancet. 1998 May 9;351(9113):1393-6. doi: 10.1016/S0140-6736(97)10384-1. PMID 9593409
- [Background] Pollak MN. Endocrine effects of IGF-I on normal and transformed breast epithelial cells: potential relevance to strategies for breast cancer treatment and prevention. Breast Cancer Res Treat. 1998 Feb;47(3):209-17. doi: 10.1023/a:1005950916707. PMID 9516077
- [Background] Wolk A, Mantzoros CS, Andersson SO, Bergstrom R, Signorello LB, Lagiou P, Adami HO, Trichopoulos D. Insulin-like growth factor 1 and prostate cancer risk: a population-based, case-control study. J Natl Cancer Inst. 1998 Jun 17;90(12):911-5. doi: 10.1093/jnci/90.12.911. PMID 9637140
- [Background] Arita Y, Kihara S, Ouchi N, Takahashi M, Maeda K, Miyagawa J, Hotta K, Shimomura I, Nakamura T, Miyaoka K, Kuriyama H, Nishida M, Yamashita S, Okubo K, Matsubara K, Muraguchi M, Ohmoto Y, Funahashi T, Matsuzawa Y. Paradoxical decrease of an adipose-specific protein, adiponectin, in obesity. Biochem Biophys Res Commun. 1999 Apr 2;257(1):79-83. doi: 10.1006/bbrc.1999.0255. PMID 10092513
- [Background] Kari FW, Dunn SE, French JE, Barrett JC. Roles for insulin-like growth factor-1 in mediating the anti-carcinogenic effects of caloric restriction. J Nutr Health Aging. 1999;3(2):92-101. PMID 10885804
- [Background] Ma J, Pollak MN, Giovannucci E, Chan JM, Tao Y, Hennekens CH, Stampfer MJ. Prospective study of colorectal cancer risk in men and plasma levels of insulin-like growth factor (IGF)-I and IGF-binding protein-3. J Natl Cancer Inst. 1999 Apr 7;91(7):620-5. doi: 10.1093/jnci/91.7.620. PMID 10203281
- [Background] Giovannucci E, Pollak MN, Platz EA, Willett WC, Stampfer MJ, Majeed N, Colditz GA, Speizer FE, Hankinson SE. A prospective study of plasma insulin-like growth factor-1 and binding protein-3 and risk of colorectal neoplasia in women. Cancer Epidemiol Biomarkers Prev. 2000 Apr;9(4):345-9. PMID 10794477
- [Background] Harman SM, Metter EJ, Blackman MR, Landis PK, Carter HB; Baltimore Longitudinal Study on Aging. Serum levels of insulin-like growth factor I (IGF-I), IGF-II, IGF-binding protein-3, and prostate-specific antigen as predictors of clinical prostate cancer. J Clin Endocrinol Metab. 2000 Nov;85(11):4258-65. doi: 10.1210/jcem.85.11.6990. PMID 11095464
- [Background] Stattin P, Bylund A, Rinaldi S, Biessy C, Dechaud H, Stenman UH, Egevad L, Riboli E, Hallmans G, Kaaks R. Plasma insulin-like growth factor-I, insulin-like growth factor-binding proteins, and prostate cancer risk: a prospective study. J Natl Cancer Inst. 2000 Dec 6;92(23):1910-7. doi: 10.1093/jnci/92.23.1910. PMID 11106682
- [Background] Amling CL, Kane CJ, Riffenburgh RH, Ward JF, Roberts JL, Lance RS, Friedrichs PA, Moul JW. Relationship between obesity and race in predicting adverse pathologic variables in patients undergoing radical prostatectomy. Urology. 2001 Nov;58(5):723-8. doi: 10.1016/s0090-4295(01)01373-5. PMID 11711349
- [Background] Berg AH, Combs TP, Du X, Brownlee M, Scherer PE. The adipocyte-secreted protein Acrp30 enhances hepatic insulin action. Nat Med. 2001 Aug;7(8):947-53. doi: 10.1038/90992. PMID 11479628
- [Background] Chang S, Hursting SD, Contois JH, Strom SS, Yamamura Y, Babaian RJ, Troncoso P, Scardino PS, Wheeler TM, Amos CI, Spitz MR. Leptin and prostate cancer. Prostate. 2001 Jan 1;46(1):62-7. doi: 10.1002/1097-0045(200101)46:13.0.co;2-v. PMID 11170133
- [Background] Hsing AW, Chua S Jr, Gao YT, Gentzschein E, Chang L, Deng J, Stanczyk FZ. Prostate cancer risk and serum levels of insulin and leptin: a population-based study. J Natl Cancer Inst. 2001 May 16;93(10):783-9. doi: 10.1093/jnci/93.10.783. PMID 11353789
- [Background] Rodriguez C, Patel AV, Calle EE, Jacobs EJ, Chao A, Thun MJ. Body mass index, height, and prostate cancer mortality in two large cohorts of adult men in the United States. Cancer Epidemiol Biomarkers Prev. 2001 Apr;10(4):345-53. PMID 11319175
- [Background] Stattin P, Soderberg S, Hallmans G, Bylund A, Kaaks R, Stenman UH, Bergh A, Olsson T. Leptin is associated with increased prostate cancer risk: a nested case-referent study. J Clin Endocrinol Metab. 2001 Mar;86(3):1341-5. doi: 10.1210/jcem.86.3.7328. PMID 11238530
- [Background] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624